CLINICAL TRIAL: NCT04471324
Title: EBUS Guided Cryobiopsies With Ultrathin Cryoprobe in Patients With Peripheral Pulmonary Nodules - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thoraxklinik-Heidelberg gGmbH (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Cryo SPN 1.1 trial
Record Dates: First submitted 2020-06-22; First posted 2020-07-15 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Transbronchial Cryobiopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EBUS cryo probe (Experimental): Patients receive a transbronchial cryobiopsy using an eBUS cryo probe
  Interventions: Device: EBUS cryo probe

INTERVENTIONS:
Device: EBUS cryo probe — patients receive a transbronchial cryo biopsy with the EBUS cryo probe from ERBE and an ultra thin bronchoskope

SUMMARY:
The standard procedure in the diagnosis of peripheral round foci is bronchoscopy with transbronchial forceps biopsy (TBB). Despite the simultaneous application of X-ray fluoroscopy, the diagnostic value of this method depends strongly on the size, location and relationship of the foci to the airways as well as their radiological representability. By inserting radial 20 MHz ultrasound probes through the working channel of a flexible bronchoscope into the periphery of the lung, the detection of peripheral foci can be improved. By simultaneously using a virtual bronchoscopy with an ultra-thin bronchoscope, even smaller round foci in the periphery of the lung can be detected. For some years now, tension-resistant cryoprobes have been used for transbronchial biopsy. Here, especially in lesions that can only be reached endoscopically tangentially, advantages have been shown over forceps biopsy. Much larger tissue samples can be obtained without increasing the complication rate. Studies showed that the combination of the EBUS navigation technique with the cryobiopsy procedure is feasible and safe in the endoscopic diagnosis of peripheral lung tumors. This study investigates to what extent the combination of an ultra-thin cryoprobe with an ultra-thin bronchoscope together with the radial EBUS can further improve the diagnosis. This study is a non-randomized pilot study to prove the feasibility of this procedure. The EBUS probe and the bronchoscope are CE certified for this application. The study will be conducted as a monocentric study at the Thorax Clinic at Heidelberg University Hospital.

A total of 30 patients with an indication for transbronchial biopsy will be prospectively included. All patients will be examined according to the clinical standard. After a freezing time of 3-7 seconds, the probe together with the bronchoscope will be extracted and the sample will be defrosted in a water-filled sample vial. Up to 4 biopsies will be taken depending on the investigator's assessment. The samples will be collected separately and the order of the biopsies will be recorded. The primary endpoint is the feasibility of the procedure. Secondary endpoints are safety, diagnostic hit rate, biopsy size and quality and success rate depending on the position of the EBUS probe (tangential or central).

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple peripheral pulmonary round foci in CT
* signed patient information

Exclusion Criteria:

* severe co-mornidity
* no signed patien information
* contraindication for intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the procedure - assessed by diagnosis agreement within the multidisciplinary team discussion | Day 1
  Pathological assessment of biopsies for ILD diagnosis

SECONDARY OUTCOMES:
Bleeding time in seconds | Day 1 until Day 2
  Assessed by using a stop watch and entering data into a questionnaire
Size of biopsies | Day 1
  Planimetry
Quality of biopsies | Day 1
  artefact-free biopsies
Exacerbation rate | 4 weeks after biopsy
  Assessment of exacerbations until 4 weeks after biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Eberhardt, Prof. Dr. med., Principal Investigator — Thoraxklinik Universitaetsklinikum Heidelberg
Locations (1):
- Thoraxklinik Universitaetsmedizin, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No